CLINICAL TRIAL: NCT00199537
Title: Bone Loss in Men on Androgen Blockade as Adjuvant Therapy for Prostate Cancer
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Lawson Health Research Institute Internal Review Fund (Unknown); University of Western Ontario, Canada (Other)
Responsible Party: Dr. Hassan Razvi, Lawson Health Research Institute
Other Study IDs: R-05-055; Lawson IRF-071-04; UWO ADF SG06-02
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Prostate Cancer; Bone Loss
MeSH Terms: conditions — Prostatic Neoplasms; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with advanced prostate cancer undergoing adjuvant treatment with androgen blockade will be followed over a 1 year interval to assess the effects of this treatment on bone metabolism. It is expected that men undergoing androgen blockade will experience accelerated bone loss.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Age of 40 years or greater
* Diagnosis of advanced prostate cancer (ie: prostate-specific antigen [PSA] less than 25 ug/L and undergoing continued treatment with leuteinizing hormone-releasing hormone [LHRH] therapy)
* Willing and able to consent

Exclusion Criteria:

* Metastatic disease to bone
* Medications affecting bone turnover (bisphosphonate, steroids, anticonvulsant)
* Renal failure (serum creatinine > 200 umol/L)
* Co-morbidity factors affecting bone density (ie: Paget's, rheumatoid arthritis)
* Factors affecting ability to perform the bone density tests using femoral head measurements (ie: bilateral hip arthroplasty)
* Cancer other than skin, except when, in the investigators' opinion, it is determined to be appropriate and not adversely affect the outcome of the trial
* Gastrointestinal (GI) pathology (eg. malabsorption syndrome)
* Parathyroid disease

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with Prostate Cancer undergoing continued treatment with leuteinizing hormone-releasing hormone [LHRH] therapy
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2005-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Razvi, MD, FRCSC, Principal Investigator — Urology, St. Joseph's Hospital, University of Western Ontario
Locations (1):
- Urology Clinic & Prostate Centre, St. Joseph's Hospital, St. Joseph's Health Care London, London, Ontario, Canada